CLINICAL TRIAL: NCT02879591
Title: Enhancing Social Interaction With an AlterEgo Artificial Agent
Acronym: ALTEREGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); Ecole Polytechnique Fédérale de Lausanne (Other); University of Bristol (Other); DEUTSCHES FORSCHUNGSZENTRUM FUER KUENSTLICHE (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: U 9038
Record Dates: First submitted 2016-07-29; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with schizophrenia (Experimental): Patients with schizophrenia
  Interventions: Other: Social Skills training with Avatar therapist
- Healthy volunteers (Placebo Comparator): Healthy volunteers
  Interventions: Other: Social Skills training with Avatar therapist

INTERVENTIONS:
Other: Social Skills training with Avatar therapist

SUMMARY:
The objective of AlterEgo is the creation of an interactive cognitive architecture, implementable in various artificial agents, allowing a continuous interaction with patients suffering from social disorders, by virtue of changes in behavioural (robot-based) as well as morphological (avatar-based) properties of that agent. The project includes research in fundamental and clinical neurosciences, interaction modeling, development of new computer-vision techniques and human-robot interfaces, as well as evaluation of the scenarios with patients before, during, and after training sessions. At the end of the project, the investigators will produce a new avatar-based clinical method able to enhance social interaction of patients.

The first challenge of this project is to create an avatar alter ego of a patient. Based on recent work in social robotics and neurosciences, the investigators hypothesize that if patients face artificial agents morphologically and behaviourally similar to them, they will increase their social interaction. The second challenge is to transform the morphology and the behaviour of the similar artificial agent into that of a healthy and different agent. The investigators assume that the smooth and continuous behavioural shift from similar/unhealthy to complementary/healthy social behaviour will lead to a better social rehabilitation. AlterEgo opens the door to a new generation of social artificial agents in service robotics. AlterEgo is an interdisciplinary project at the interaction of Social Motor Neurosciences (UM1), Robotics (EPFL), Complex Systems Dynamics (UOB), Computer Vision (DFKI), and Psychiatry (CHU).

This project includes a set of experiments that started in april 2014 and will terminate in september 2016 before undergoing a randomised clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from schizophrenia according to the criteria proposed in the DSM-IV-TR
* Aged between 18 and 60 years old.

Exclusion Criteria:

* History of head trauma
* History of neurological disorders (epilepsy disease, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Huntington's disease, stroke)
* An actual ECT treatment
* Substance Abuse and / or current Substance dependence (excluding tobacco and cannabis).
* Pregnant women, new mothers and nursing mothers
* People private of their liberty

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 246 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
number of patient enhancing social intercation | 3 months
  improvement of social interactions (interpersonal relations, items 1 to 7 on Specific Levels Of Functioning, SLOF)

SECONDARY OUTCOMES:
number of patient accepting avatar therapy | 3 months
questionnaire for Faisability of avatar therapy | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service Universitaire de psychiatrie adulte, University Hospital of Montpellier, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No